CLINICAL TRIAL: NCT03202147
Title: A Phase II Safety and Efficacy Study of ALZT-OP1a as Adjuvant Treatment in Subjects With Post-Ischemic Stroke Cognitive Impairment (PSCI)
Brief Title: Safety and Efficacy of ALZT-OP1a as Adjuvant Treatment in Subjects With Post-Ischemic Stroke Cognitive Impairment (PSCI)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely prior to initiation but potentially will resume in the future.
Sponsor: AZTherapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZT-003
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2020-04

CONDITIONS: Ischemic Stroke; Post-stroke Cognitive Impairment
Keywords: Ischemic stroke, post-stroke cognitive impairment, PSCI
MeSH Terms: conditions — Ischemic Stroke | interventions — Cromolyn Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALZT-OP1a (Active Comparator): ALZT-OP1a: cromolyn (17.1 mg, capsule) for oral inhalation via dry powder inhaler, taken twice per day (morning and evening), 8-12 hours apart.
  Interventions: Drug: Cromolyn
- Placebo (Placebo Comparator): ALZT-OP1a: placebo capsule for oral inhalation via dry powder inhaler, taken twice per day (morning and evening), 8-12 hours apart.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cromolyn — Active capsules for inhalation.
  Other Names: Cromolyn sodium
  Arms: ALZT-OP1a
Other: Placebo — Non-active capsules for inhalation.
  Arms: Placebo

SUMMARY:
This is a Phase II, randomized, double-blinded, placebo-controlled study for subjects with evidence of PSCI.

DETAILED DESCRIPTION:
This Phase II study is designed as a randomized, double-blinded, placebo-controlled study for subjects with evidence of PSCI.

Subjects will be randomly assigned to the Group I arm (ALZT-OP1a adjuvant treatment), which will consist of ALZT-OP1a for inhalation, taken twice daily (morning and evening), OR the Group II placebo arm, which will consist of inhaled placebo, taken twice daily (morning and evening).

A minimum of 350 subjects will be randomized to receive one of two possible treatment assignments: ALZT-OP1a adjuvant treatment of active study drug or placebo.

To account for subject dropouts (estimated rate of 30%), it is anticipated that up to 500 (or 250 subjects per treatment arm) may be recruited and randomized, to achieve a minimum of 175 evaluable subjects per treatment arm.

Randomization assignments will be stratified by site to ensure balance by site.

ELIGIBILITY:
Inclusion Criteria

* Male or female, aged 18 years or above;
* Subject has suffered a recent (within 1-7 days) ischemic stroke supported by CT scan or MRI findings;
* Subject has a score on the NIHSS of 5-14 (inclusive);
* Evidence of stroke related cognitive impairment, documented by neuropsychological evaluation and a Clinical Dementia Rating (Global) ≥ 0.5;
* Must be fluent in the language of the cognitive testing material being administered;
* Study partner is available who has frequent contact with the participant (e.g. an average of 10 hours per week or more), and can accompany the participant to all clinic visits for the duration of the protocol;
* Visual and auditory acuity adequate for neuropsychological testing.

Exclusion Criteria:

* Subject has medical history of dementia (prior to current ischemic stroke event);
* Subject has a known medical history of major depression or psychotic disorder;
* Unstable cardiovascular or cerebrovascular disease;
* Aphasia or other disability severe enough to prevent valid neuropsychiatric assessment;
* History of any other significant neurological disease prior to ischemic stroke;
* History of schizophrenia or bipolar disorder (DSM-IV criteria);
* History of alcohol or substance abuse or dependence within the past 3 years (DSM-IV criteria);
* Currently taking medications that could lead to difficulty complying with the protocol;
* Investigational agents are prohibited one month prior to entry and for the duration of the trial;
* Currently taking cromolyn, or has taken cromolyn, within the past 12 months;
* Allergy to cromolyn (also known as Intal®, Nasalcrom®, Opticrom®, Gastrocrom®, etc.);
* Clinically significant respiratory disorders with impaired respiratory effort or difficulty taking inhaled drugs (examples: Stage III-IV chronic obstructive pulmonary disease [COPD], emphysema);
* Uncontrolled chronic asthma;
* Taking inhaled protein products on a chronic basis (such as insulin, parathyroid hormone [PTH], etc.);
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol;
* Pregnancy or lactation for female subjects of child-bearing potential (i.e., < two years post-menopausal or not surgically sterile);
* For sexually active male subjects, unwillingness or incapability of using appropriate contraception methods;
* Severe renal or hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline and Week 12
  The primary endpoint is the difference in performance in the ALZT-OP1a adjuvant treatment group compared to the placebo group, as quantified by the mean change from baseline to Week 12 scored on MoCA.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline and Week 12
  The secondary endpoint is the difference in performance in the ALZT-OP1a adjuvant treatment group compared to the placebo group, as quantified by the mean change from baseline to week 12 in points scored on MMSE.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Brazier, BS, Study Director — AZTherapies, Inc.

IPD SHARING:
Plan to Share IPD: No